CLINICAL TRIAL: NCT06314828
Title: A Phase 1, Open-label, Single Arm Clinical Trial to Evaluate the Tolerability, Safety and Efficacy of RJMty19 in Subjects With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: A Tolerability, Safety and Efficacy Study of RJMty19 in Subjects With Relapsed or Refractory B-NHL
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Ruishun Biotech Co., Ltd (Industry)
Collaborators: Ruijin Hospital (Other); Southern Medical University, China (Other); Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJMty19-B-NHL002
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-01

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: off-the-shelf cell product; CAR-DNT; Cell Therapy; B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RJMty19 (CD19-CAR-DNT Cells) (Experimental): The trial is divided into two parts: Part A is a dose escalation trial with four dose groups (5×10^6 CAR+ cells/kg, 1×10^7 CAR+ cells/kg, 2×10^7 CAR+ cells/kg and 4×10^7 CAR+ cells/kg at day 0), with 8-24 patients planned to be enrolled. Part B is a dose-expansion trial in which 3~6 patients will receive RJMty19 infusions at RP2D dose levels.
  Interventions: Biological: RJMty19 (CD19-CAR-DNT cells)

INTERVENTIONS:
Biological: RJMty19 (CD19-CAR-DNT cells) — Lentiviral vector-transducted double negative T cells (DNT) to express anti-CD19 CAR. Prior to cellular infusion, each patient received cyclophosphamide, fludarabine and Etoposide lymphodepleting chemotherapy.

SUMMARY:
This is a Phase 1, open-label, single-arm study to evaluate tolerability, safety and efficacy of RJMty19 in adult subjects with r/r B-NHL.

DETAILED DESCRIPTION:
The study was based on an accelerated titration and "3+3" design with a dose-escalation phase and a dose-expansion phase, and was designed to assess the safety, maximum tolerated dose, pharmacokinetic profile, and initial efficacy of RJMty19 in subjects with r/r B-NHL after second-line treatment or above.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the subsequent follow-up.
2. Aged 18 to 65 years (including cut-offs), regardless of gender.
3. B-cell non-Hodgkin's lymphoma diagnosed as CD19-positive by cytology or histopathology according to WHO 2022 criteria, including pathologically confirmed (1) diffuse large B-cell lymphoma, non-specific type (DLBCL, NOS); (2) follicular lymphoma histopathologically graded as grade 3b (FL3b); (3) follicular lymphoma with diffuse large B-cell transformation; (4) primary mediastinal large B-cell lymphoma (PMBCL); (5) high-grade B-cell lymphoma (HGBCL).
4. Relapsed/refractory B-cell non-Hodgkin's lymphoma, provided one of the following conditions is met:

   1. Definition of relapse: Relapse after achieving remission (PR and CR) with second-line or higher therapy;
   2. Definition of refractory:

      * No response to second-line or more therapy: The best efficacy of last therapy is PD or SD (SD requires at least 2 cycles of treatment);
      * Recurrence (must have biopsy-proven recurrence) or progression within 12 months of autologous stem cell transplantation (ASCT) . If salvage therapy, no response to last therapy (SD or PD).
5. Subjects must have received adequate treatment in the past, which should include the following treatments:

   1. Anti-CD20 monoclonal antibody, unless the investigator determines that the tumor is CD20 negative;
   2. Chemotherapy containing anthracycline drugs;
   3. For subjects with transformed follicular lymphoma (tFL) who have been previously treated with follicular lymphoma (FL) chemotherapy and with transformation to DLBCL show refractory to chemotherapy.
6. ECOG performance status 0 to 1.
7. The presence of a measurable lesion that meets one of the following criteria:

   1. The long axis of the lymph node lesion exceeds 15 mm in length (the short axis is measurable);
   2. The long and short axes of the extralymph node lesion exceed 10 mm in length.
8. ALaboratory results within 7 days prior to Lymphodepletion need to meet the following criteria:

   1. Coagulation function:

      * Activated partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN);
      * Prothrombin time (PT) ≤ 1.5 times ULN;
   2. Liver function:

      * Glutathione aminotransferase (AST) ≤ 5 times the upper limit of normal (ULN);
      * Glutamic aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN);
      * Total bilirubin ≤ 1.5 times ULN, unless the subject has documented Gilbert syndrome;
      * Subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included.
   3. Renal function:

      * Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min;
   4. Complete blood count (No blood transfusion treatment received within 7 days prior to examination):

      * Haemoglobin ≥ 80 g/L;
      * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L;
      * A platelet count ≥ 50 x 10^9/L;
   5. Cardiopulmonary function:

      * Left ventricular ejection fraction (LVEF) ≥ 45%;
      * Oxygen saturation ≥ 91%;
9. Female subjects with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female subjects of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female subjects without childbearing potential (meeting at least 1 of the following criteria) is described below:

   1. Have undergone a hysterectomy or bilateral oophorectomy;
   2. Medically recognised ovarian failure;
   3. Medically recognised as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).

Exclusion Criteria:

1. Other malignancies within 5 years prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, post-radical localized prostate cancer, post-radical ductal carcinoma in situ, and post-radical thyroid cancer
2. Any unstable systemic disease: including but not limited to active infection (other than local infection), unstable angina, cerebrovascular accident or transient ischaemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (refractory hypertension is defined as blood pressure that has not reached standard after >1 month of reasonably tolerable treatment with ≥3 antihypertensive drugs (including diuretics) at adequate doses based on lifestyle improvement or blood pressure that is not effectively controlled with ≥4 antihypertensive drugs), severe cardiac arrhythmias requiring pharmacologic treatment, hepatic arrhythmias, liver diseases, kidney diseases or metabolic disorders.
3. Patients with B-cell non-Hodgkin's lymphoma with active central nervous system invasion.
4. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titres not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA ,positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test.
5. Subjects who are receiving systemic steroids prior to screening and who are judged by the investigator to require long-term treatment with systemic steroids during the treatment period (except for inhaled or topical use).
6. Previous organ transplantation or preparation for organ transplantation (except for haematopoietic stem cell transplantation).
7. Persons with acute/chronic Graft-vs-Host Disease (GvHD).
8. Patients have received a haematopoietic stem cell transplant within 2 months prior to screening.
9. Active neurological autoimmune or inflammatory diseases (e.g. Guillain-Barre Syndrome (GBS), Amyotrophic lateral sclerosis (ALS)).
10. Clinically significant active cerebrovascular diseases (such as cerebral edema, posterior reversible encephalopathy syndrome).
11. Patients with a life expectancy of less than 3 months.
12. Subjects have participated in other interventional clinical studies within 3 months prior to screening.
13. Received attenuated live vaccine within 6 weeks prior to lymphodepletion.
14. The subjects have contraindications or hypersensitivity reactions to fludarabine, cyclophosphamide, etoposide, tocilizumab, investigational product and its ingredients.
15. Remaining within the washout period of other antitumor treatments prior to lymphodepletion.
16. Patients who, in the investigator's judgment and/or clinical criteria, have a contraindication to any of the study procedures or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of RJMty19 for R/R B-NHL subjects
Maximum Tolerated Dose (MTD) | Up to 28 days
  MTD is the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 90 days
  The peak concentration of CD19-CAR-DNT cells amplified in the peripheral blood (Cmax, detected by qPCR and Flow Cytometry).
Pharmacokinetics (PK) indicator (AUC) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by qPCR and Flow Cytometry).
Pharmacokinetics (PK) indicator (Tmax) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the peak plasma time (Tmax). Tmax is defined as the time to reach the highest concentration (Tmax, detected by qPCR and Flow Cytometry).
Pharmacokinetics (PK) indicator (T1/2) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of CD19-CAR-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by qPCR and Flow Cytometry).
Overall Response Rate | Up to 2 years
  The proportion of CR or PR patients as assessed by investigators based on Lugano 2014 Response Assessment
Disease Control Rate | Up to 2 years
  The percentage of PR, CR and SD patients in the total patient population
Duration of Response | Up to 2 years
  The time from the start of the first assessment of CR or PR to the first assessment as disease recurrence or progression or death
Progression Free Survival | Up to 2 years
  The length of time that a participant's disease did not progress during or after RJMty19 infusion.
Overall Survival | Up to 15 years
  From the date of entry into the clinical study until death from any cause
Overall Response Rate at 3 months | Up to 3 months
  The percentage of PR and CR patients in the total patient population at 3 months